CLINICAL TRIAL: NCT06647446
Title: Improvements in Function and Pain in the Rehabilitation of Patients with Knee Osteoarthritis Using an Exercise Program Telemonitored Compared to Conventional Treatment
Acronym: KNEE_Telemon
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rodrigo Martín-San-Agustin, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3407154
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise supported by the digital physiotherapy and telerehabilitation software TRAK (Experimental): Home therapeutic exercise intervention scheduled through the software of digital physiotherapy and telerehabilitation TRAK
  Interventions: Other: Exercise supported by the digital physiotherapy and telerehabilitation software TRAK
- Standard home-based exercise (Active Comparator): Home therapeutic exercise program scheduled through a dossier and an exercise diary
  Interventions: Other: Standard home-based exercise

INTERVENTIONS:
Other: Exercise supported by the digital physiotherapy and telerehabilitation software TRAK — 8 week home therapeutic exercise program that includes flexibility and strength exercises scheduled through the software of digital physiotherapy and telerehabilitation TRAK. The program will be carried out with a frequency of 3 weekly sessions, preferably on alternate days. The program will be carried out with the support of the TRAK software (https://www.trakphysio.com/es/), which allows the exercises to be carried out in front of a camera that, with the help of an artificial intelligence system, offers feedback to the participant and allows you to keep a record of the sessions. As an addition to the home sessions, two face-to-face sessions will be held in the first and fifth weeks, respectively. The exercise program includes three levels of difficulty (easy, intermediate and difficult), with patients advancing to subsequent levels once each level is successfully overcome.
  Arms: Exercise supported by the digital physiotherapy and telerehabilitation software TRAK
Other: Standard home-based exercise — 8 week home therapeutic exercise program that includes flexibility and strength exercises scheduled through a dossier and an exercise diary. The program will be carried out with a frequency of 3 weekly sessions, preferably on alternate days. The program will be carried out with the support of an information dossier of the exercises to be performed and a monitoring diary in which everything related to the sessions carried out will be noted.. As an addition to the home sessions, two face-to-face sessions will be held in the first and fifth weeks, respectively. The exercise program includes three levels of difficulty (easy, intermediate and difficult), with patients advancing to subsequent levels once each level is successfully overcome.
  Arms: Standard home-based exercise

SUMMARY:
Osteoarthritis is a very prevalent pathology after the fifth decade of life. It usually appears in the hip and hand, although its presence in the knee is even greater, with a prevalence in subjects over 45 years of age of 19% radiographically (radiographic findings without taking symptoms into account) and 7% in the symptomatic population, for those over 60 years of age, 37% radiographic and 12% symptomatic and finally, for those over 75 years of age there was 50% of osteoarthritis of the knee diagnosed by radiographs and 33% were symptomatic. There are gender differences: the lifetime risk of suffering knee osteoarthritis is estimated at 40% for men and 47% for women. Furthermore, the impact of this pathology is significant, being the most frequent cause of gait-related disability in adults in the United States.

Different approaches have been proposed for the treatment of knee osteoarthritis. Currently, clinical practice guidelines place therapeutic exercise and education as the first line of treatment, reserving joint replacement surgery in case of failure of conservative treatment and only if there is severe disability.

In recent years, due to the pandemic, there has been an accelerated development of telemedicine and telerehabilitation in all its aspects. Applications and websites have been developed for online rehabilitation. An example of this is TRAK, a telerehabilitation web tool that allows the creation of a profile for each patient and the design of personalized exercise programs and the periodization of the sessions to be carried out. During the execution of the exercises, the screen of the split phone will appear, displaying on one side the execution of the exercise by a model and on the other side, the patient sees himself performing the exercise. This tool allows the monitoring of the therapeutic exercise without the need to go to a consultation or to be in front of a physiotherapist, reducing the economic and time investment.

Thus, the present work tries to compare the treatment with exercises monitored by means of the TRAK application with the performance of the same exercises, without the help of this tool.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with osteoarthritis of the knee.
* Age >45 years.
* The patient presents with knee pain during physical activity.
* The patient reports knee symptoms in the last month.
* The patient has a mobile phone with internet access.

Exclusion Criteria:

* Previous knee surgeries.
* Planned surgeries during the duration of the trial.
* Patient is currently undergoing physical therapy.
* Patient currently has severe pathology that may compromise participation in the exercise program (advanced COPD, cardiac or arterial disease).
* Associated rheumatic pathology (fibromyalgia, gout, rheumatoid arthritis).
* BMI >30.
* Having completed a strengthening exercise program in the last year.
* Visual disturbances that prevent being able to observe the cell phone screen correctly.
* Lack of digital skills in the use of the Internet with the cell phone.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disability | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Disability measured using the scale Western Ontario and Mc Caster Universities Osteoarthritis (WOMAC) which consists in a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright.
Pain | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Numeric Rating Scale (NRS-11); the 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
40 metre fast-paced walk | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Tests short distance walking ability with changing direction. A timed walk of 4 x 10 metres for a total of 40 metres.
30 seconds chair-stand test | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand. While monitoring the participant's performance to ensure proper form, the tester silently counts the completion of each correct stand.
Kinesiphobia | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Kinesiofobia measured using the Tampa Scale of Kinesiofobia (range score from 17 [lower levels of kinesiophobia]-68 [higher levels of kinesiophobia])
Medication intake | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Medication intake registered using a diary
Adherence | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Adherence measured using the TRAK application
Adherence | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Adherence measured using an exercise diary